CLINICAL TRIAL: NCT05269667
Title: SAkuraBonsai: Clinical, Imaging And Biomarker Open-Label Study In Neuromyelitis Optica Spectrum Disorder (NMOSD) With Satralizumab As An Intervention
Brief Title: A Study In Neuromyelitis Optica Spectrum Disorder (NMOSD) With Satralizumab As An Intervention
Acronym: SAkuraBonsai
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study has proved infeasible to recruit in sufficient numbers. There are insufficient eligible patients presenting to sites.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical Co. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MN42928; 2021-001088-26 (EudraCT Number)
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Neuromyelitis Optica Spectrum Disorder; NMOSD
MeSH Terms: conditions — Neuromyelitis Optica | interventions — satralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: treatment-naïve NMOSD patients (Experimental): Patients will be treated with 120 mg satralizumab subcutaneously (SC) as monotherapy at Weeks 0, 2 (±3 days), 4 (±3 days), and then every 4 weeks (±3 days) till the last administration at Week 92 followed by a clinical evaluation at Week 96. The first dose at Week 0 (baseline visit) will be administered at the study site by the designated site staff during the scheduled study visit. All assessments (clinical, laboratory and imaging) should be performed before satralizumab administration. The next dose at Week 2 will be self-administered by the patient under the supervision of a designated study staff at the study site. All the subsequent doses will be self-administered by the patient following training from a healthcare provider (for patients who are not able to administer satralizumab SC by themselves, support by a caregiver/nurse is advised).
  Interventions: Drug: Satralizumab 120 mg
- Cohort 2: NMOSD patients who are inadequate responders to previous treatment with RTX (Experimental): Patients will be treated with 120 mg satralizumab subcutaneously (SC) as monotherapy at Weeks 0, 2 (±3 days), 4 (±3 days), and then every 4 weeks (±3 days) till the last administration at Week 92 followed by a clinical evaluation at Week 96. The first dose at Week 0 (baseline visit) will be administered at the study site by the designated site staff during the scheduled study visit. All assessments (clinical, laboratory and imaging) should be performed before satralizumab administration. The next dose at Week 2 will be self-administered by the patient under the supervision of a designated study staff at the study site. All the subsequent doses will be self-administered by the patient following training from a healthcare provider (for patients who are not able to administer satralizumab SC by themselves, support by a caregiver/nurse is advised).
  Interventions: Drug: Satralizumab 120 mg

INTERVENTIONS:
Drug: Satralizumab 120 mg — Satralizumab 120 mg will be administered as monotherapy (SC) in the abdominal or femoral region at Weeks 0, 2 (±3 days), 4 (±3 days), and then every 4 weeks (±3 days) till the last administration at Week 92 followed by a clinical evaluation at Week 96. The first dose at Weeks 0 (baseline visit) will be administered at the study site by the designated site staff during the scheduled study visit. The next dose at Week 2 will be self-administered by the patient under the supervision of a designated study staff at the study site. All the subsequent doses will be self-administered by the patient following training from a healthcare provider (for patients who are not able to administer satralizumab SC by themselves, support by a caregiver/nurse is advised).

SUMMARY:
Objective of the trial is to describe the efficacy and safety of satralizumab in patients with aquaporin-4 (AQP4) antibody seropositive NMOSD, either treatment naive or inadequate responders to previous treatment with rituximab (RTX) (or its biosimilar)

DETAILED DESCRIPTION:
Neuromyelitis optica (NMO) and neuromyelitis optica spectrum disorder (NMOSD) are severe demyelinating inflammatory autoimmune neurological disorders. The estimated global pooled prevalence of NMOSD is 1.82 per 100 000 people (Etemadifar et al. 2015). The disorder is characterized by inflammatory lesions in the optic nerve, spinal cord, brainstem, and cerebrum; and clinically by optic neuritis (ON) and/or transverse myelitis causing potentially severe motor and sensory impairment, bladder dysfunction, vision loss, pain, and other debilitating symptoms (Wingerchuk et al. 2015). Recovery is variable, and inflammatory attacks often result in permanent disability. Untreated, the risks of severe disability or death are substantial (Jarius et al. 2014).

NMOSD is radiologically and prognostically distinct from multiple sclerosis (MS), and has a pathophysiology unresponsive to typical MS treatment (Weinshenker 2007; Oh, and Levy et al. 2012).

ELIGIBILITY:
Inclusion criteria

* Age 18 to 74 years, inclusive, at the time of informed consent
* Have a diagnosis of AQP4 antibody seropositive NMOSD according to the International Panel for NMO Diagnosis (IPND) criteria
* For women of childbearing potential: agreement to either remain abstinent (refrain from heterosexual intercourse) or to use reliable means of contraception (physical barrier [patient or partner] in conjunction with a spermicidal product, contraceptive pill, patch, injectables, intrauterine device or intrauterine system) during the treatment period and for at least 3 months after the last dose of study drug Cohort 1 (treatment-naïve NMOSD patients)
* Confirmation of NMOSD diagnosis with AQP4+ antibodies
* Have clinical evidence of at least 1 documented attack or relapse (including first attack) in the last year prior to screening
* Naive to maintenance therapy (disease-modifying therapy [DMT] or immunosuppressive therapy [IST]) Cohort 2 (NMOSD patients with inadequate response to RTX [or its biosimilar])
* Confirmation of NMOSD diagnosis and AQP4+ antibodies in the disease history of the patient
* Have a length of disease duration from first symptom of ≤5 years
* History of ongoing treatment with RTX (or its biosimilar) (at least 2 infusions) for NMOSD with a maximum duration of 6 months since last administration prior to enrolment in the study
* Ongoing disease activity after last RTX (or its biosimilar) infusion i.e., relapse and/or any new inflammatory event, confirmed by magnetic resonance imaging (MRI) or ophthalmological assessment

Exclusion criteria Exclusion criteria for both the cohorts

* Inability to complete an MRI
* Participants who are pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final dose of satralizumab
* Any surgical procedure (except for minor surgeries) within 4 weeks prior to baseline
* Evidence of other demyelinating disease, including MS or progressive multifocal leukoencephalopathy (PML)
* Evidence of serious uncontrolled concomitant diseases that may preclude patient participation
* Active or presence of recurrent bacterial, viral, fungal, mycobacterial infection or other infection (excluding fungal infections of nail beds or caries dentium) at baseline
* Infection requiring hospitalization or treatment with intravenous (IV) anti-infective agents within 4 weeks prior to baseline visit
* Evidence of chronic active hepatitis B
* Evidence of active tuberculosis (TB)
* History or laboratory evidence of coagulation disorders
* Receipt of a live or live-attenuated vaccine within 6 weeks prior to baseline
* Presence or history of malignancy
* History of drug or alcohol abuse within 1 year prior to baseline
* History of diverticulitis that, in the Investigator's opinion, may lead to increased risk of complications such as lower gastrointestinal perforation
* History of severe allergic reaction to a biologic agent
* Active suicidal ideation within 6 months prior to screening, or history of suicide attempt within 3 years prior to screening
* Treatment with any investigational agent within 6 months prior to baseline or 5 drug elimination half-lives of the investigational agent (whichever is longer) Cohort 1 (treatment-naïve NMOSD patients)
* Any previous treatment with IL-6 inhibitory therapy (e.g., tocilizumab), alemtuzumab, total body irradiation, stem-cell therapy, or bone marrow transplantation
* Any previous treatment with eculizumab, belimumab, natalizumab, glatiramer acetate, fingolimod, teriflunomide, dimethyl fumarate, siponimod, or ozanimod
* Any previous treatment with anti-CD4, cladribine or mitoxantrone
* Any previous treatment with B-cell depleting agents
* Any previous treatment with immunosuppressants Cohort 2 (NMOSD patients with inadequate response to RTX)
* Discontinued RTX (or biosimilar) treatment due to any other reason than inadequate response to treatment

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- University of Kansas Medical Center, Kansas City, Kansas, United States
- National Cancer Center, Goyang-si, South Korea
- Ondokuz Mayis University School of Medicine, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 3 investigative sites in 3 countries.
Pre-assignment Details: A total of 4 participants with neuromyelitis optica spectrum disorder (NMOSD) were enrolled in 'Cohort 2: Inadequate Responders to Previous Rituximab (RTX) Treatment' to receive satralizumab. No participants were enrolled in 'Cohort 1: Treatment-naïve Participants' due to early study termination.
Groups:
- Cohort 2: Inadequate Responders to Previous Rituximab (RTX) Treatment: Participants with inadequate response to previous RTX treatment received 120 mg of satralizumab monotherapy as SC injection on Day 1 of Weeks 0, 2, 4 and then Q4W up to Week 92.
Period: Overall Study
Arm/Group | Cohort 2: Inadequate Responders to Previous Rituximab (RTX) Treatment
Started | 4
Completed | 0
Not Completed | 4
Not completed — Study Terminated by Sponsor | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants who received any dose of satralizumab.
Groups:
- Cohort 2: Inadequate Responders to Previous RTX Treatment: Participants with inadequate response to previous RTX treatment received 120 mg of satralizumab monotherapy as SC injection on Day 1 of Weeks 0, 2, 4 and then Q4W up to Week 92.
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Relapse-Free Participants
Description: Relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur <31 days following the onset of a relapse were considered part of the same relapse.
Time Frame: Up to 14 months
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
percentage of participants | 100

2. Primary Outcome: Annualized Relapse Rate (ARR)
Description: The ARR was calculated descriptively by dividing the total number of relapses for all participants by the total years of drug exposure. Relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur <31 days following the onset of a relapse were considered part of the same relapse.
Time Frame: Up to 14 months
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Number (95% Confidence Interval); unit: relapses per participant-year
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
relapses per participant-year | 0 [0 to 0]

3. Primary Outcome: Time to First Relapse (TFR)
Description: TFR was defined as the time from first dose of satralizumab to the first occurrence of relapse. Relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur <31 days following the onset of a relapse were considered part of the same relapse.
Time Frame: Up to 14 months
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
weeks | NA [NA to NA] — Median and 95% Confidence Interval (CI) was not estimable due to no participants with events.

4. Primary Outcome: Percentage of Participants Hospitalized Due to Relapse
Description: Relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur <31 days following the onset of a relapse were considered part of the same relapse. The severity of relapses was assessed based on the occurrence of hospitalization.
Time Frame: Up to 14 months
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
percentage of participants | 0

5. Primary Outcome: Percentage of Participants Using Corticosteroids Due to Relapse
Description: Relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur <31 days following the onset of a relapse were considered part of the same relapse. The severity of relapses was assessed based on use of corticosteroids.
Time Frame: Up to 14 months
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
percentage of participants | 0

6. Primary Outcome: Percentage of Participants in Need of Rescue Therapy Due to Relapse
Description: Relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur <31 days following the onset of a relapse were considered part of the same relapse. The severity of relapses was assessed based on the need of rescue therapy. Rescue therapy for clinical relapse included pulse intravenous (IV) corticosteroids, oral corticosteroids for tapering, intravenous immunoglobulin (IVIG) and/or apheresis (including plasma exchange and plasmapheresis).
Time Frame: Up to 14 months
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
percentage of participants | 0

7. Primary Outcome: Percentage of Participants in Need of Plasma Exchange Due to Relapse
Description: Relapse was the occurrence of new or worsening neurological symptoms attributable to NMOSD. New or worsening neurological symptoms that occur <31 days following the onset of a relapse were considered part of the same relapse. The severity of relapses was assessed based on the need for plasma exchange.
Time Frame: Up to 14 months
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
percentage of participants | 0

8. Primary Outcome: Percentage of Participants With Residual Disability Due to Relapse
Description: as for outcome 1
Time Frame: Up to 14 months
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
percentage of participants | 0

9. Primary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Score
Description: EDSS was a quantitative measure of disability and for assessment of severity of relapse for participants with NMOSD. The overall score ranges from 0 points (normal neurological examination) up to 10 points (death), increasing in increments of 0.5 points. Higher scores represent increased disability. A negative change from baseline indicates improvement.
Time Frame: Up to Week 36
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
score on a scale | 0 (0)

10. Primary Outcome: Time to Onset of Confirmed Disability Progression (CDP) Sustained for at Least 12 Weeks
Description: EDSS was a quantitative measure of disability and for assessment of severity of relapse for participants with NMOSD. The overall score ranges from 0 points (normal neurological examination) up to 10 points (death), increasing in increments of 0.5 points. Higher scores represent increased disability. CDP was defined as 1-point or greater worsening in EDSS from baseline that is not attributable to another etiology when the baseline score is 5.5 or less, and ≥ 0.5 when the baseline score is above 5.5. Disability progression was considered confirmed when the increase in the EDSS is confirmed at a regularly scheduled visit at least 12 weeks after the initial documentation of neurological worsening.
Time Frame: Up to 12 weeks
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
weeks | NA [NA to NA] — Median and 95% CI were not estimable due to no participants with events.

11. Primary Outcome: Change From Baseline in the Symbol Digital Modalities Test (SDMT)
Description: SDMT testing was to detect impairment of key neurocognitive functions that underlie many substitution tasks, including sustained attention, visual scanning, and recent memory. The test consisted of a sequence of 110 symbols displayed in a maximum 90 seconds and a reference key legend with 9 symbols in a given order and their respective matching digits from 1 to 9. The test measures the speed (number of correct paired responses) to pair abstract symbols with specific digits in 90 seconds time. The score is the number of correctly paired items in 90 seconds with a maximum score of 110 and minimum of 0. Higher scores indicate improvement.
Time Frame: Baseline, Week 24
Population: ITT population included all enrolled participants who received any dose of satralizumab. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 1
score on a scale | -5 (NA) — The standard deviation (SD) was not estimable as only a single participant was evaluable.

12. Primary Outcome: Change in High Contrast (100%) and Low Contrast (2.5%) Visual Acuity Using High-and Low-contrast Letter Acuity (LCLA) Charts
Description: Best corrected high-contrast (100%) and low-contrast (2.5%) visual acuities were measured at distances of both 4 and 1 meters with the appropriate eye charts. Each eye was tested individually. No visual acuities were obtained with both eyes open. The participants read the charts from left to right starting with the top line (largest letters). The participants proceeded to each lower line until he/she could not see the letters. The total number of letters read correctly were recorded for each eye. Visual acuity was measured before any drops are instilled into the eye and before OCT assessments.
Time Frame: Baseline and Week 24
Population: as for outcome 11
Measure: Number; unit: Letters correct
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 1
Letters correct
  Right High Contrast | -14
  Left High Contrast | 80
  Right Low Contrast | 60
  Left Low Contrast | 33

13. Primary Outcome: Change in Visual Functioning Questionnaire -25 (VFQ-25)
Description: The National Eye institute (NEI) VFQ-25 captures a participants's perception of vision-related functioning and vision-related quality of life. The core measures include 25 items that comprise 11 vision-related subscales and one item on general health. The NEI VFQ-25 also included an appendix of additional items that was used to expand the scales up to 39 total items. The composite score and the subscale scores range from 0 to 100, with higher scores indicating better vision-related functioning.
Time Frame: At Week 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 1
score on a scale | 10 (NA) — The SD was not estimable as only a single participant was evaluable.

14. Secondary Outcome: Count of T2-weighted Fluid-Attenuated Inversion-Recovery (FLAIR) Hyperintense Lesions Assessed Using Magnetic Resonance Imaging (MRI) Scans
Description: MRI was used to monitor central nervous system (CNS) lesions and potentially other pathophysiology, such as inflammation and neurodegeneration. LETM=longitudinally extensive transverse myelitis. Stm=subcortical temporal medial. Count of T2-weighted FLAIR hyperintense lesions (including new and enlarging) were distributed across the following regions: cerebrum, optic nerves, optic chiasm, area postrema, brainstem and cerebellum.
Time Frame: Weeks 4, 8, 12 and 24
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Number; unit: number of lesions
Units Other Than Participants: lesion
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
Number analyzed (lesion) | 9
number of lesions
  Baseline: Hyperintense Lesion: number analyzed (lesion) | 3
  Baseline: Hyperintense Lesion | 3
  Week 4: Hyperintense Lesion: number analyzed (lesion) | 3
  Week 4: Hyperintense Lesion | 3
  Week 8: Hyperintense Lesion: number analyzed (lesion) | 3
  Week 8: Hyperintense Lesion | 2
  Week 12: Hyperintense Lesion: number analyzed (lesion) | 3
  Week 12: Hyperintense Lesion | 3
  Baseline: Hyperintense Letm Lesion: number analyzed (lesion) | 2
  Baseline: Hyperintense Letm Lesion | 2
  Week 4: Hyperintense Letm Lesion: number analyzed (lesion) | 2
  Week 4: Hyperintense Letm Lesion | 2
  Week 8: Hyperintense Letm Lesion: number analyzed (lesion) | 2
  Week 8: Hyperintense Letm Lesion | 1
  Week 12: Hyperintense Letm Lesion: number analyzed (lesion) | 2
  Week 12: Hyperintense Letm Lesion | 1
  Baseline: Hyperintense Stm Lesion | 9
  Week 4: Hyperintense Stm Lesion | 8
  Week 8: Hyperintense Stm Lesion | 8
  Week 12: Hyperintense Stm Lesion | 8
  Week 24: Hyperintense Lesion: number analyzed (lesion) | 3
  Week 24: Hyperintense Lesion | 1
  Week 24: Hyperintense Letm Lesion: number analyzed (lesion) | 2
  Week 24: Hyperintense Letm Lesion | 0
  Week 24: Hyperintense Stm Lesion | 1

15. Secondary Outcome: Volume of T2-weighted FLAIR Hyperintense Lesions Assessed Using MRI Scans
Description: MRI was used to monitor CNS lesions and potentially other pathophysiology, such as inflammation and neurodegeneration.
Time Frame: Baseline, Week 12
Population: as for outcome 11
Measure: Median (Standard Deviation); unit: milliliter (mL)
Units Other Than Participants: lesion
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 1
Number analyzed (lesion) | 1
milliliter (mL)
  Baseline | 0.2285 (NA) — The SD was not estimable as only a single participant was evaluable.
  Week 12 | 0.2520 (NA) — The SD was not estimable as only a single participant was evaluable.

16. Secondary Outcome: Number of Participants With Contrast-enhancing T1-weighted Lesions (CEL) Assessed Using MRI Scans
Description: MRI was used to monitor CNS lesions and potentially other pathophysiology, such as inflammation and neurodegeneration.
Time Frame: Basline, Weeks 4, and 12
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
Participants | 0

17. Secondary Outcome: Number of Participants With Diffusion Abnormalities, Microbleeds and Cerebral Perfusion Alterations Assessed Using MRI Scans
Time Frame: Up to 14 Months
Population: Data for this outcome measure was not collected and analyzed as planned as the study was terminated per sponsor's decision.
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

18. Secondary Outcome: Number of Participants With Global and Regional Brain Volume Loss Assessed Using MRI Scans
Time Frame: Up to 14 Months
Population: as for outcome 17
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

19. Secondary Outcome: Number of Participants With New and Persisting Short T1 Inversion Recovery (STIR)/ Proton Density (PD) Hyperintense Lesions and T1-weighted Contrast Enhancement Assessed Using MRI Scans
Time Frame: Up to 14 months
Population: as for outcome 17
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

20. Secondary Outcome: Quantitative T1 Mapping (Magnetization Prepared Rapid Gradient Echo Sequence [MP2RAGE]) Assessed Using MRI Scans
Time Frame: Up to 14 months
Population: as for outcome 17
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

21. Secondary Outcome: T2*/R* Ratio for Iron Concentration Estimation Assessed Using MRI Scans
Time Frame: Up to 14 months
Population: as for outcome 17
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

22. Secondary Outcome: Quantitative Diffusion/ Diffusion Tensor Imaging (DTI) Assessed Using MRI Scans
Time Frame: Up to 14 months
Population: as for outcome 17
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

23. Secondary Outcome: Change in the Retinal Nerve Fiber Layer (RNFL) Thickness Assessed Using Optical Coherence Tomography (OCT)
Time Frame: Up to 14 months
Population: as for outcome 17
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

24. Secondary Outcome: Change in the Ganglion Cell Plus Inner Plexiform (GCIP) Layer Thickness Assessed Using OCT
Time Frame: Up to 14 months
Population: as for outcome 17
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

25. Secondary Outcome: Concentration of Satralizumab in Cerebrospinal Fluid (CSF) and Serum
Time Frame: Baseline and Week 12
Population: ITT population included all enrolled participants who received any dose of satralizumab. Data for this CSF concentartion was not collected and analyzed as planned as the study was terminated per sponsor's decision.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/litre (ng/L)
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
nanograms/litre (ng/L) | 19078.02 (15.94)

26. Secondary Outcome: Number of Participants With Anti-satralizumab Antibodies
Time Frame: Up to 14 months
Population: as for outcome 17
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 0

27. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. A SAE is any significant hazard, contraindication, side effect that is fatal or life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is medically significant or requires intervention to prevent one or other of the outcomes listed above. An AESI included drug induced liver injury and suspected transmission of infectious agent via medicinal products.
Time Frame: Up to 14 months
Population: Safety population included all enrolled participants who received any dose of satralizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
Participants
  AE | 2
  SAE | 0
  AESIs | 0

28. Primary Outcome: Time to Onset of Confirmed Disability Progression (CDP) Sustained for at Least 24 Weeks
Description: as for outcome 10
Time Frame: Up to 24 weeks
Population: ITT population included all enrolled participants who received any dose of satralizumab.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
Number analyzed (Participants) | 4
weeks | NA [NA to NA] — Median and 95% CI was not estimable due to no participants with events.

ADVERSE EVENTS:
Time Frame: Up to 14 months
Description: Safety population included all enrolled participants who received any dose of satralizumab.
Arm/Group | Cohort 2: Inadequate Responders to Previous RTX Treatment
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 2: Inadequate Responders to Previous RTX Treatment (N=4)
Injection site reaction (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigators are free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT05269667/Prot_SAP_000.pdf